CLINICAL TRIAL: NCT00351936
Title: A Placebo-Controlled, Cross-Over Trial of Aripiprazole Added to Obese Olanzapine-Treated Patients With Schizophrenia
Brief Title: A Placebo-Controlled, Cross-Over Trial of Aripiprazole
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North Suffolk Mental Health Association (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, David C. Henderson, MD, Associate Professor of Psychiatry, Harvard University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-2005
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Diabetes; Obesity; Olanzapine; Insulin Resistance
MeSH Terms: conditions — Schizophrenia; Diabetes Mellitus; Obesity; Insulin Resistance | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aripiprazole (Active Comparator): aripiprazole 15mg/day
  Interventions: Drug: Aripiprazole
- placebo (Placebo Comparator): matched placebo for aripiprazole 15mg/day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Aripiprazole
  Arms: Aripiprazole
Drug: placebo
  Arms: placebo

SUMMARY:
This study is a ten-week, placebo-controlled, double-blind, cross-over, randomized trial of the novel antipsychotic agent, aripiprazole, added to 20 obese stable olanzapine-treated patients with schizophrenia or schizoaffective disorder. The advantage of the crossover design is that each subject will act as their own control and fewer subjects will be required than a between-group design.

DETAILED DESCRIPTION:
Specific Aims:

This study is a ten-week, placebo-controlled, double-blind, cross-over, randomized trial of the novel antipsychotic agent, aripiprazole, added to 20 obese stable olanzapine-treated patients with schizophrenia or schizoaffective disorder. The advantage of the crossover design is that each subject will act as their own control and fewer subjects will be required.

Study Procedures:

We have designed this trial to examine effects upon weight, lipids, glucose metabolism, positive symptoms, negative symptoms, and depressive symptoms. This project, examining the usefulness of combination therapy, may offer a possible intervention for patients who are obese and treated with olanzapine, but otherwise experiencing a good clinical response. Many patients, despite the medical problems that may occur, are reluctant to switch their antipsychotic agent.

Location:

This study will be performed at the Freedom Trail Clinic of the Erich Lindemann Mental Health Center by faculty of the Schizophrenia Program of the Massachusetts General Hospital and staff of the Freedom Trail Clinic.

Subjects:

Subjects will include 20 stable outpatients with schizophrenia or schizoaffective disorder treated with olanzapine for at least one year. Prior to enrollment, we will determine that the clinician has optimized the dose of the antipsychotic and maintained the medication at a stable dose for at least 1 month. Patients will be excluded for significant medical illness, substance abuse, or inability to provide informed consent.

Safety Assessments:

Medication Trial:

Patients will have a baseline assessment performed and then randomized to placebo or aripiprazole 15 mg/day for 4 weeks. After the initial 4 weeks of medication patients will be reassessed, have a 2-week washout period and then crossover to the other treatment for another 4 weeks. The olanzapine dose will be unchanged during the trial. Patients will be given a two-week supply of medication at baseline and week 2 and then again at weeks 6 and 8.

Screening Visit The diagnosis of schizophrenia or schizoaffective disorder will be confirmed by a research psychiatrist using DSM IV criteria. A physical examination will be performed and medical history, vital signs, weight, height, waist/hip circumference, skin-fold measurements, 12-lead EKG and demographic information will be obtained. Laboratory measures will include olanzapine blood levels, fasting glucose, insulin, basic chemistry profiles, liver enzymes, CBC, lipid profile, leptin, LDL- particle size, PAI-1, C-reactive protein, sICAM, vWF and a DNA sample will be drawn at screening for future analysis of the 5-HT-2C and H1 receptor genes.

Baseline Assessment:

The following scales will be completed at baseline and will comprise the treatment efficacy battery: Positive and Negative Syndrome Scale (PANSS), Scale for Assessment of Negative Symptoms (SANS), Clinical Global Impressions scale (CGI), Hamilton Depression Rating Scale (HAM-D), Global Assessment Scale (GAS), Fatigue Scale Inventory (FSI) Trauma History Questionnaire (THQ) and the Quality of Life Scale (QOL). A single rater will perform all assessments. If it is necessary to use a second rater, inter-rater reliability will be established before the addition of the second rater and will be repeated every three months by use of videotaped interviews. The treatment efficacy battery will be repeated at week 4, 6 and 10 except for the THQ, which will only be administered at the beginning of the study.

Safety and Monitoring Assessments:

Blood pressure, heart rate, temperature, weight, waist/hip circumference will be performed at each visit (baseline, weeks 2, 4, 6, 8 and 10). Side effects will be monitored at baseline and weeks 2, 4, 6, 8, and 10 using the Systematic Assessment for Treatment Emergent Events (SAFTEE). Body fat composition will be measured by skin-fold calipers at baseline, week 4, 6 and 10. EPS will be evaluated at baseline and weeks 2, 4, 6, 8 and 10 using the Simpson-Angus Scale, Barnes Akathisia Scale, and the Abnormal Involuntary Movement Scale (AIMS).

Measure of Energy Expenditure and Dietary Assessment:

Patients will be asked to wear an accelerometer for four consecutive days to obtain an objective measure of physical activity. During the same four days the patients will maintain a four-day food record of all food and beverages consumed. This will provide a means of assessing energy intake verses energy output. Patients will also complete the Modifiable Activity Questionnaire (MAQ). Energy expenditure and dietary intake will be assessed at baseline, weeks 4, 6 and 10.

Randomization:

The double-blind, placebo-controlled, crossover study will consist of two random order 4-week treatment arms (aripiprazole 15 mg or placebo) separated by a 2-week adjuvant treatment washout. Following baseline, subjects will be randomized, double-blind, to either aripiprazole or placebo for 4 weeks. After the initial 4 weeks of medication patients will be reassessed, have a 2-week washout period and then crossover to the other treatment for another 4 weeks.

Subject Recruitment:

Potential subjects will be identified by their clinicians at the Freedom Trail Clinic. Patients will give their physician verbal permission to be contacted for research purposes. A member of the research team will meet with the subject and explain the study protocol, including a review of risks and potential benefits. A copy of the study consent form will be provided to the patient at this time. Patients who express interest after this first meeting will be evaluated for competency to provide informed consent by a physician who is not a member of the research team. Patients who are judged to be competent will then be asked to meet with the principal investigator who will review the study protocol and consent form with the patient and obtain informed consent. The human rights officer of the North Suffolk Mental Health Association will be asked to participate in this meeting unless the patient declines. Family and residential staff will also be invited to participate if the patient agrees.

Potential Risks:

Aripiprazole did not produce any serious adverse effects in animal and human safety studies. No consistent abnormality of vital signs, laboratory, EKG or EEG has emerged. In clinical trials, no side effects occurred at rates greater than 2x placebo. Nausea, vomiting, anxiety, headache, dyspepsia, somnolence, orthostatic hypotension, tachycardia, insomnia, akathisia, EPS, and weight gain may be potential side effects.

Benefits:

It is not known if aripiprazole added to olanzapine will help a subject's mood, motivation, hallucinations, and unusual experiences. Other patients may benefit if this study finds that aripiprazole added to olanzapine is useful for treating symptoms of schizophrenia.

Data Management and Statistical Analysis:

Data management and statistical analysis will be provided by Dr. David Schoenfeld from the Massachusetts General Hospital, Biostatistics Center.

Protection of Human Subjects:

Principal members of our research team have all completed certification for protection of human subjects in clinical trials. The clinical protocol will be submitted for approval by the institutional review boards of the Massachusetts Department of Mental Health. Potential subjects will be referred by their clinicians. Clinicians will be asked to sign a statement that verifies that the patient is interested in participating, understands that participation is voluntary, and understands that declining participation will not affect treatment at the facility. A member of the research team will meet with the patient and explain the study protocol, including a review of risks and potential benefits. A copy of the study consent form will be provided to the patient at that time to share with family members or residential staff. Patients who continue to express interest after this first meeting will be evaluated by a physician who is not a member of the research team for capacity to provide informed consent. Patients who are judged to be competent will then be asked to meet with the principal investigator or co-investigator who will review the study protocol and consent form with the patient and obtain informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18-65
* Diagnosis of schizophrenia, any subtype, or schizoaffective disorder, any sub-type
* Body mass index > 30 Kg/m2 or >27 Kg/m2 with other risk factors (HTN, Lipid abnormalities)
* Well established compliance with outpatient medications.
* Maintained on a stable dose of olanzapine for at least one month.

Exclusion Criteria:

* Serious medical or neurological illness (unstable cardiac disease, malignancy, liver or renal impairment, etc.)
* Current substance abuse
* Psychiatrically unstable, which is defined as a score on the CGI's severity of illness question of 5 or greater or a baseline Total PANSS score > 75
* Pregnancy, nursing, or unwilling to use appropriate birth control measures during participation if female and fertile
* Serious suicidal or homicidal risk within the past three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Henderson, MD, Principal Investigator — North Suffolk Mental Health Association
Locations (1):
- Freedom Trail Clinic, Boston, Massachusetts, United States

REFERENCES:
- [Background] Allison DB, Mentore JL, Heo M, Chandler LP, Cappelleri JC, Infante MC, Weiden PJ. Antipsychotic-induced weight gain: a comprehensive research synthesis. Am J Psychiatry. 1999 Nov;156(11):1686-96. doi: 10.1176/ajp.156.11.1686. PMID 10553730
- [Background] Baptista T, Beaulieu S. Body weight gain, insulin, and leptin in olanzapine-treated patients. J Clin Psychiatry. 2001 Nov;62(11):902-4. doi: 10.4088/jcp.v62n1111b. No abstract available. PMID 11775052
- [Background] Beasley CM Jr, Hamilton SH, Crawford AM, Dellva MA, Tollefson GD, Tran PV, Blin O, Beuzen JN. Olanzapine versus haloperidol: acute phase results of the international double-blind olanzapine trial. Eur Neuropsychopharmacol. 1997 May;7(2):125-37. doi: 10.1016/s0924-977x(96)00392-6. PMID 9169300
- [Background] Beasley CM Jr, Tollefson GD, Tran PV. Safety of olanzapine. J Clin Psychiatry. 1997;58 Suppl 10:13-7. PMID 9265911
- [Background] Davis JM, Chen N, Glick ID. A meta-analysis of the efficacy of second-generation antipsychotics. Arch Gen Psychiatry. 2003 Jun;60(6):553-64. doi: 10.1001/archpsyc.60.6.553. PMID 12796218
- [Background] Gupta S, Droney T, Al-Samarrai S, Keller P, Frank B. Olanzapine: weight gain and therapeutic efficacy. J Clin Psychopharmacol. 1999 Jun;19(3):273-5. doi: 10.1097/00004714-199906000-00014. No abstract available. PMID 10350036
- [Background] Henderson DC, Kunkel L, Nguyen DD, Borba CP, Daley TB, Louie PM, Freudenreich O, Cather C, Evins AE, Goff DC. An exploratory open-label trial of aripiprazole as an adjuvant to clozapine therapy in chronic schizophrenia. Acta Psychiatr Scand. 2006 Feb;113(2):142-7. doi: 10.1111/j.1600-0447.2005.00612.x. PMID 16423166
- [Background] Kay SR, Opler LA, Lindenmayer JP. Reliability and validity of the positive and negative syndrome scale for schizophrenics. Psychiatry Res. 1988 Jan;23(1):99-110. doi: 10.1016/0165-1781(88)90038-8. PMID 3363019
- [Background] Levine J, Schooler NR. SAFTEE: a technique for the systematic assessment of side effects in clinical trials. Psychopharmacol Bull. 1986;22(2):343-81. No abstract available. PMID 3774930
- [Background] Osser DN, Najarian DM, Dufresne RL. Olanzapine increases weight and serum triglyceride levels. J Clin Psychiatry. 1999 Nov;60(11):767-70. doi: 10.4088/jcp.v60n1109. PMID 10584766
- [Background] Pi-Sunyer FX. Medical hazards of obesity. Ann Intern Med. 1993 Oct 1;119(7 Pt 2):655-60. doi: 10.7326/0003-4819-119-7_part_2-199310011-00006. PMID 8363192
- [Background] Pi-Sunyer FX. The medical risks of obesity. Obes Surg. 2002 Apr;12 Suppl 1:6S-11S. doi: 10.1007/BF03342140. PMID 11969107
- [Background] Wirshing DA, Wirshing WC, Kysar L, Berisford MA, Goldstein D, Pashdag J, Mintz J, Marder SR. Novel antipsychotics: comparison of weight gain liabilities. J Clin Psychiatry. 1999 Jun;60(6):358-63. PMID 10401912

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects will be identified by their clinicians at the Freedom Trail Clinic. Targeted enrollment will include 20 stable outpatients with schizophrenia or schizoaffective disorder treated with olanzapine for at least one year. Patients will be excluded for significant medical illness, and substance abuse.
Pre-assignment Details: Sixteen subjects consented to participate. One subject was found ineligible for the study due to recent changes in medications and did not reach baseline/group assignment. Available data from the remaining 15 subjects are included in all analyses.
Groups:
- Cross-over Aripiprazole and Placebo: This double-blind, placebo-controlled, crossover study consisted of 2 random-order 4-week treatment arms(aripiprazole 15 mg or placebo) separated by a 2-week adjuvant treatment washout. After baseline, subjects were randomized, double blind, to either aripiprazole or placebo for 4 weeks. After the initial 4 weeks of medication, subjects were reassessed, had a 2-week washout period, and then another complete assessment before receiving the other treatment of another 4 weeks. All assessments were again repeated at week 10.
Period: Overall Study
Arm/Group | Cross-over Aripiprazole and Placebo
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cross-over Aripiprazole and Placebo
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49.87 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weight (Lbs)
Description: Evaluating change in weight (lbs) between Baseline and Week 4, comparing subjects treated with aripiprazole for 4 weeks to subjects treated with placebo for 4 weeks.
Time Frame: baseline, week 4
Measure: Mean (Standard Deviation); unit: lbs
Groups:
- Aripiprazole: Olanzapine-treated subjects took adjunctive aripiprazole 15mg/day tablets for 4 weeks.
- Placebo: Olanzapine-treated subjects took adjunctive placebo tablets (to match aripiprazole 15mg/day tablets) for 4 weeks.
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 15 | 15
lbs | -2.9 (4.7) | 2.1 (3.3)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA

2. Primary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Evaluating change in Body Mass Index (BMI) between Baseline and Week 4, comparing subjects treated with aripiprazole for 4 weeks to subjects treated with placebo for 4 weeks.
Time Frame: baseline, week 4
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 15 | 15
kg/m^2 | -0.4 (0.7) | 0.3 (0.5)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA

3. Primary Outcome: Change From Baseline in Waist-hip Ratio (WHR)
Description: Evaluating change in waist-hip ratio (WHR) between Baseline and Week 4, comparing subjects treated with aripiprazole for 4 weeks to subjects treated with placebo for 4 weeks.
Time Frame: baseline, week 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 15 | 15
cm | 0.0 (0.0) | 0.0 (0.0)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Superiority or Other; p = 0.747, ANCOVA

4. Primary Outcome: Change From Baseline in Fasting Total Cholesterol
Description: Evaluating change in fasting total cholesterol between Baseline and Week 4, comparing subjects treated with aripiprazole for 4 weeks to subjects treated with placebo for 4 weeks.
Time Frame: baseline, week 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 15 | 15
mg/dL | -3 (24) | 9 (22)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Superiority or Other; p = 0.208, ANCOVA

5. Primary Outcome: Change From Baseline in Low-density Lipoprotein (LDL)
Description: Evaluating change in low-density lipoprotein (LDL) between Baseline and Week 4, comparing subjects treated with aripiprazole for 4 weeks to subjects treated with placebo for 4 weeks.
Time Frame: baseline, week 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 15 | 15
mg/dL | -0.2 (22.2) | 3.1 (15)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Superiority or Other; p = 0.665, ANCOVA

6. Primary Outcome: Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C)
Description: Evaluating change in high-density lipoprotein cholesterol (HDL-C) between Baseline and Week 4, comparing subjects treated with aripiprazole for 4 weeks to subjects treated with placebo for 4 weeks.
Time Frame: baseline, week 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 15 | 15
mg/dL | 0.4 (7.2) | 0.6 (3.0)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Superiority or Other; p = 0.999, ANCOVA

7. Primary Outcome: Change From Baseline in Triglycerides
Description: Evaluating change in triglyceride levels between Baseline and Week 4, comparing subjects treated with aripiprazole for 4 weeks to subjects treated with placebo for 4 weeks.
Time Frame: baseline, week 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 15 | 15
mg/dL | -51.7 (78.2) | 47.6 (52.7)
Statistical Analysis 1: Comparison: Aripiprazole vs Placebo; Test type: Superiority or Other; p = 0.001, ANCOVA

ADVERSE EVENTS:
Arm/Group | Cross-over Aripiprazole and Placebo
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cross-over Aripiprazole and Placebo (N=15)
diarrhea (Gastrointestinal disorders) | 1 (1) — At the time of the event, subject was in her 2-week washout phase of the study, therefore not on any study medication. Subject has a history of chronic diarrhea and takes antidiarrheal medications as needed.

LIMITATIONS AND CAVEATS:
The small sample size and the short duration of active treatment and washout period may have prevented detection of other metabolic benefits, including possible reductions in fasting insulin and insulin resistance (measured by HOMA-IR).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes